CLINICAL TRIAL: NCT04599686
Title: Androgen Deprivation Therapy (ADT) Versus Stereotactic Body Radiotherapy (SBRT) for Oligometastatic Prostate Cancer: A Prospective Randomized Control Clinical Trial
Brief Title: Stereotactic Body Radiotherapy (SBRT) for Oligometastatic Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Changhai Ho
Record Dates: First submitted 2020-10-10; First posted 2020-10-23 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-12

CONDITIONS: Treatment
Keywords: SBRT; Oligometastatic Prostate Cancer; Feasibility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADT (Active Comparator): Evaluating men with oligometastatic prostate cancer lesions randomized to ADT.
  Interventions: Drug: ADT
- SBRT (Experimental): Evaluating men with oligometastatic prostate cancer lesions randomized to stereotactic body radiation therapy (SBRT).
  Interventions: Radiation: SBRT

INTERVENTIONS:
Drug: ADT — On the day of enrollment, luteinizing hormone-releasing hormone agonist (LHRHa) was given for ADT.
  Arms: ADT
Radiation: SBRT — Evaluating men with oligometastatic prostate cancer lesions randomized to stereotactic body radiation therapy (SBRT) (3-5 fractions).
  Arms: SBRT

SUMMARY:
The aim of this study is to test the safety and feasibility of SBRT without ADT in oligometastatic prostate cancer in patients for whom the standard treatment is ADT, and to further explore how long only radiotherapy for oligometastases can prolong biochemical progression-free survival (bPFS). In this study, men with oligometastatic prostate cancer lesions will be randomized (1:1) to ADT versus SBRT. Within 6 weeks of the oligometastases diagnosis, ADT or SBRT (30-50Gy with 3-5 fractions) will be administered.

DETAILED DESCRIPTION:
The oligometastatic disease state is an increasingly recognized phenomenon in prostate cancer. Ga-68 PSMA PET/CT has high accuracy in the diagnosis metastases from prostate cancer. In this protocol, pretreatment Ga-68 PSMA PET/ CT shall be performed in all patients.

ADT is considered standard of care treatment for advanced prostate cancer. But hormonal therapy can have side effects that greatly trouble men and lead to castration-resistant prostate cancer (CRPC). Any effort to delay the start of hormonal therapy would be an advantage to the patient. Stereotactic body radiation therapy (SBRT) is highly focused radiation, given in a very dose intensive fashion and delivered in usually less than one week. SBRT has been shown to be very effective on bone or lymph nodes metastases. Therefore, we are studying the safety and feasibility of SBRT on patients with five or fewer prostate cancer bone or lymph nodes metastases to determine if we can stall the use of hormonal therapy and/or prevent other site metastases from developing elsewhere in the body.

ELIGIBILITY:
Inclusion Criteria:

* 80 years old

  * Histologically confirmed adenocarcinoma of the prostate
  * Prostate cancer treated with curative intent (radical prostatectomy, primary radiotherapy, or a combination of both)
  * Ga-68 prostate-specific membrane antigen (PSMA) PET/CT evidence of one to three metastases (bone or lymph node) within 6 weeks of enrolment, if the position of oligometastases is judged by the doctor to be in the same radiotherapy area, the number of metastases can be appropriately increased to 5
  * Without ADT treatment
  * PSA< 50ng/ml
  * ECOG performance status 0-2
  * Written informed consent according to ICH/GCP regulations before registration and prior to any trial specific procedures

Exclusion Criteria:

* Any previous or ongoing treatment of oligometastases including radiotherapy, ADT, chemotherapy, focal treatment, etc.
* Unstable lesions with spinal or long bone metastases
* A tumor located at less than 3 mm from the urethra or rectum when measured at the MRI

  * 4 metastases, or if the metastases are in the same radiotherapy area, ≥6 metastases
* Histologically confirmed neuroendocrine tumor or small cell carcinoma of the prostate
* Severe or active co-morbidity likely to impact on the advisability of SBRT like severe liver or kidney dysfunction, etc.
* Patients with other malignancies, or acute or other severe infections, with ulcerative colitis, inflammatory bowel disease, etc.
* Patients who have participated in other clinical trials for less than three months
* Unsuitable to participate in this clinical trial judged by the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-11 (Estimated); Primary Completion 2022-11-11 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
1-year ADT-free survival of the experimental group | Assessment ADT-free survival of the experimental group at 1 year
  To assess ADT-free survival of the experimental group
The Probability of Radiotherapy-related Toxicity | Assessment Toxicity at 1 year
  Radiotherapy-related complications
The time from inception of the study to castration-resistant prostate cancer (CRPC) | Assessment at 1 year
  the time from inception of the study to castration-resistant prostate cancer (CRPC)

SECONDARY OUTCOMES:
1-year Efficacy Biochemical Progression-free Survival (bPFS) | 1 year
  Biochemical Progression-free Survival (bPFS)
1-year Local Progression-Free-Survival(LPFS) | Assessment at 1 year
  Local Progression-Free-Survival(LPFS)
1-year Distant Metastasis Free Survival(DMFS) | Assessment at 1 year
  Distant Metastasis Free Survival(DMFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including baseline characteristics,treatment information and follow-up data on toxicity, survival and disease control will be shared.
Supporting Information: Study Protocol
Time Frame: Within 5 years after the publication of the study.
Access Criteria: Data may be shared with radiation oncologists who are interested in examining the efficacy and toxicity of oligometastatic prostate cancer treated with stereotactic body radiotherapy (SBRT) or androgen deprivation therapy (ADT). Detailed study protocol should be emailed along with the request of the data. We may carefully review the study protocol, and data will only be shared with well-designed studies.
URL: http://clinicaltrials.gov/ct2/show/NCT04599686?term=NCT04599686&draw=2&rank=1

REFERENCES:
- [Derived] Zhao X, Wang T, Ye Y, Li J, Gao X, Zhang H. Stereotactic body radiotherapy (SBRT) versus androgen deprivation therapy (ADT) for oligometastatic prostate cancer: protocol for a prospective randomised control clinical trial. BMJ Open. 2022 Sep 30;12(9):e051371. doi: 10.1136/bmjopen-2021-051371. PMID 36180115
- Available data/document: Study Protocol: NCT04599686 — http://clinicaltrials.gov/ct2/results?cond=&term=NCT04599686&cntry=&state=&city=&dist= — Please see the clinical trials NCT04599686